CLINICAL TRIAL: NCT01993108
Title: Control of Cognition: Naltrexone, Methylphenidate, and ADHD Study
Brief Title: Control of Cognition (Naltrexone, Methylphenidate, and ADHD Study (NMAS))
Acronym: NMAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Chandra Sekhar Sripada, Assistant Professor of Psychiatry at the University of Michigan, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HUM00047129
Record Dates: First submitted 2013-11-13; First posted 2013-11-25 (Estimated); Results first posted 2018-06-18 (Actual); Last update posted 2018-06-18 (Actual); Status verified 2018-05

CONDITIONS: Healthy; Attention Deficit Hyperactivity Disorder
Keywords: Methylphenidate; Naltrexone; Placebo; Neuroimaging; Prefrontal Control Circuits; Attention Control; Motor Control; Appetitive Control
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate; Naltrexone; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Healthy Controls (Experimental): Healthy individuals will receive a one-time, randomized dose of 40mgs of Methylphenidate, 40mgs of Naltrexone, and a placebo one hour before the fMRI scanning session.
  Interventions: Drug: Methylphenidate; Drug: Naltrexone; Drug: Placebo
- Adult Attention-Deficit/Hyperactivity Disorder (Experimental): ADHD individuals will receive a one-time, randomized dose of 40mgs of Methylphenidate, 40mgs of Naltrexone, and a placebo one hour before the fMRI scanning session.
  Interventions: Drug: Methylphenidate; Drug: Naltrexone; Drug: Placebo

INTERVENTIONS:
Drug: Methylphenidate — One dose 40mgs of methylphenidate one hour before fMRI scanning.
  Other Names: Ritalin
Drug: Naltrexone — One dose 40mgs of naltrexone one hour before fMRI scanning.
  Other Names: ReVia
Drug: Placebo — One dose of placebo one hour before fMRI scanning.
  Other Names: sugar pill

SUMMARY:
The goal of this research is to understand the functioning of 'regulatory circuits' in the brain. We are also interested in how the medications methylphenidate and naltrexone affect these regulatory circuits. This research study will use a scanning technique known as functional magnetic resonance imaging (fMRI) which takes a special kind of picture of the brain that enables us to "see the brain at work". Adult participants will be given a one-time dose of either methylphenidate, naltrexone,or placebo before each fMRI scan session.

The main purpose for this research is to better understand the functioning of regulatory circuits in healthy individuals and individuals with psychiatric disorders. This research may one day help us develop better treatments for these disorders.

DETAILED DESCRIPTION:
The goal of this research is to understand the functioning of 'regulatory circuits' in the brain. These are brain circuits which allow a person to regulate their attention, regulate their behavioral responses, and regulate their decision-making. We are also interested in how the medications methylphenidate and naltrexone affect these regulatory circuits. Methylphenidate is a widely-used, FDA approved medication used to treat Attention Deficit Hyperactivity Disorder (ADHD) and is also known as Ritalin. Naltrexone is an FDA approved medication used to help treat alcohol and substance abuse.

This research study will use a scanning technique known as functional magnetic resonance imaging (fMRI)which takes a special kind of picture of the brain that enables us to "see the brain at work". Adult participants will be given a one-time dose of either methylphenidate, naltrexone,or placebo before each fMRI scan session. There are three total fMRI scan sessions. Therefore, each participant will receive each possible medication/placebo only once.

Using the fMRI technique, the main purpose of this research is to better understand the functioning of regulatory circuits in healthy individuals and individuals with psychiatric disorders. This research may one day help us develop better treatments for these disorders.

ELIGIBILITY:
Inclusion Criteria for all study participants:

* Right-Handedness

Exclusion Criteria for all study participants:

* Any clinically significant history of cardiac problems
* Any current Axis I psychiatric diagnosis as verified by the Structured Clinical Interview for DSM-IV (other than participants with ADHD or history of alcohol dependence)
* A previous adequate trial with methylphenidate (Ritalin) or naltrexone (ReVia)
* Currently taking any psychoactive medications
* Any clinically significant medical condition
* Any clinically significant neurological problem (seizures, tics, serious head injury)
* Contraindications to MRI (metal objects in body or claustrophobia)
* Currently pregnant or lactating
* Alcohol or substance abuse (current or in the past 2 years)
* Left-handedness or ambidextrous
* Liver or kidney disease

Inclusion Criteria for the participants with ADHD:

* Currently un-medicated adults with ADHD
* Has met full DSM-IV-R criteria (at least six of nine symptoms)for inattentive or hyperactive/impulsive subtypes (or both) by age 7 as well within the past month
* Has described a chronic course of ADHD symptomatology from childhood to adulthood
* Has endorsed a moderate or severe level of impairment attributed to the ADHD symptoms

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandra Sekhar Sripada, MD, PhD, Principal Investigator — University of Michigan
Locations (1):
- Rachel Upjohn Building, East Medical Campus, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Controls | Adult Attention-Deficit/Hyperactivity Disorder
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Controls | Adult Attention-Deficit/Hyperactivity Disorder | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 12 | 23
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.9 (5.0) | 22.08 (3.4) | 23.4 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 7 | 8 | 15
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Reaction Time Variability on the Multi-Source Interference Task
Description: Multi-Source Interference Task is a psychological task that measures the psychological construct of cognitive control, the ability to suppress automatic response tendencies. Reaction time variability is the standard deviation of the trial to trial reaction time measured in seconds.
Time Frame: 2 hours
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Methlyphenidate in Healthy Controls: 40mg methylphenidate in Healthy Controls
- Naltrexone in Healthy Controls: 40mg Naltrexone in Healthy Controls
- Placebo in Healthy Controls: Placebo Pill in Healthy Controls
- Methlyphenidate in ADHD: 40mg methylphenidate in ADHD
- Naltrexone in ADHD: 40mg naltrexone in ADHD
- Placebo in ADHD: Placebo Pill in ADHD
Arm/Group | Methlyphenidate in Healthy Controls | Naltrexone in Healthy Controls | Placebo in Healthy Controls | Methlyphenidate in ADHD | Naltrexone in ADHD | Placebo in ADHD
Number analyzed (Participants) | 11 | 11 | 11 | 12 | 12 | 12
seconds | .22 (.07) | .23 (.06) | .26 (.06) | .20 (.06) | .20 (.05) | .21 (.06)
Statistical Analysis 1: Comparison: Methlyphenidate in Healthy Controls vs Placebo in Healthy Controls; Test type: Superiority; p = .02, t-test, 2 sided; Mean Difference (Final Values) = 0.03
Statistical Analysis 2: Comparison: Naltrexone in Healthy Controls vs Placebo in Healthy Controls; Test type: Superiority; p = .118, t-test, 2 sided; Mean Difference (Final Values) = .02
Statistical Analysis 3: Comparison: Methlyphenidate in ADHD vs Placebo in ADHD; Test type: Superiority; p = .349, t-test, 2 sided; Median Difference (Final Values) = .02
Statistical Analysis 4: Comparison: Naltrexone in ADHD vs Placebo in ADHD; Test type: Superiority; p = .348, t-test, 2 sided; Median Difference (Final Values) = .02

2. Secondary Outcome: Reaction Time on the Multi-Source Interference Task
Description: Reaction time of the Multi-Source Interference Task is measured in seconds.
Time Frame: Two hours
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Methlyphenidate in Healthy Controls | Naltrexone in Healthy Controls | Placebo in Healthy Controls | Methlyphenidate in ADHD | Naltrexone in ADHD | Placebo in ADHD
Number analyzed (Participants) | 11 | 11 | 11 | 12 | 12 | 12
seconds | .78 (.12) | .83 (.10) | .85 (.14) | .71 (.10) | .73 (.09) | .77 (.10)
Statistical Analysis 1: Comparison: Methlyphenidate in Healthy Controls vs Placebo in Healthy Controls; Test type: Superiority; p = .019, t-test, 2 sided; Mean Difference (Final Values) = .07
Statistical Analysis 2: Comparison: Naltrexone in Healthy Controls vs Placebo in Healthy Controls; Test type: Superiority; p = .240, t-test, 2 sided; Mean Difference (Final Values) = .02
Statistical Analysis 3: Comparison: Methlyphenidate in ADHD vs Placebo in ADHD; Test type: Superiority; p = .081, t-test, 2 sided; Median Difference (Final Values) = .06
Statistical Analysis 4: Comparison: Naltrexone in ADHD vs Placebo in ADHD; Test type: Superiority; p = .247, t-test, 2 sided; Median Difference (Final Values) = .04

3. Secondary Outcome: Accuracy on the Multi-Source Interference Task
Description: Accuracy is the calculated percentage of correct responses over total trials in the Multi-Source Interference Task.
Time Frame: Two hours
Measure: Mean (Standard Deviation); unit: percent of total trials
Groups:
- Methlyphenidate in ADHD: 40mg methlyphenidate in ADHD
Arm/Group | Methlyphenidate in Healthy Controls | Naltrexone in Healthy Controls | Placebo in Healthy Controls | Methlyphenidate in ADHD | Naltrexone in ADHD | Placebo in ADHD
Number analyzed (Participants) | 11 | 11 | 11 | 12 | 12 | 12
percent of total trials | 96 (2) | 93 (7) | 91 (8) | 93 (10) | 93 (8) | 92 (5)
Statistical Analysis 1: Comparison: Methlyphenidate in Healthy Controls vs Placebo in Healthy Controls; Test type: Superiority; p = .049, t-test, 2 sided; Mean Difference (Final Values) = .05
Statistical Analysis 2: Comparison: Naltrexone in Healthy Controls vs Placebo in Healthy Controls; Test type: Superiority; p = .497, t-test, 2 sided; Mean Difference (Final Values) = .02
Statistical Analysis 3: Comparison: Methlyphenidate in ADHD vs Placebo in ADHD; Test type: Superiority; p = .814, t-test, 2 sided; Mean Difference (Final Values) = 0
Statistical Analysis 4: Comparison: Naltrexone in ADHD vs Placebo in ADHD; Test type: Superiority; p = .593, t-test, 2 sided; Mean Difference (Net) = .01

4. Secondary Outcome: Characterize the Effects of Methylphenidate and Naltrexone on Neural Circuits in Prefrontal Cortex Associated With Top-down Control.
Description: The effects of methylphenidate, naltrexone, and placebo on the change in BOLD (Blood Oxygen Level Dependent) signal will be characterized in the incongruent condition (cognitive regulation condition) of the MSIT (multi-source interference task) relative to the congruent condition (no regulation condition). Specifically, the summed BOLD signal in three regions--dorsal lateral prefrontal cortex, anterior insula, anterior cingulate--are measured.
Time Frame: Two hours
Measure: Mean (Standard Deviation); unit: Mean percentage of BOLD signal change
Arm/Group | Methlyphenidate in Healthy Controls | Naltrexone in Healthy Controls | Placebo in Healthy Controls | Methlyphenidate in ADHD | Naltrexone in ADHD | Placebo in ADHD
Number analyzed (Participants) | 11 | 11 | 11 | 12 | 12 | 12
Mean percentage of BOLD signal change | .21 (.51) | .51 (.58) | .20 (.45) | .43 (.40) | .58 (.59) | .47 (.56)
Statistical Analysis 1: Comparison: Methlyphenidate in Healthy Controls vs Placebo in Healthy Controls; Test type: Superiority; p = .926, t-test, 2 sided; Mean Difference (Final Values) = .01
Statistical Analysis 2: Comparison: Naltrexone in Healthy Controls vs Placebo in Healthy Controls; Test type: Superiority; p = .126, t-test, 2 sided; Mean Difference (Final Values) = .31
Statistical Analysis 3: Comparison: Methlyphenidate in ADHD vs Placebo in ADHD; Test type: Superiority; p = .852, t-test, 2 sided; Mean Difference (Final Values) = .04
Statistical Analysis 4: Comparison: Naltrexone in ADHD vs Placebo in ADHD; Test type: Superiority; p = .552, t-test, 2 sided; Median Difference (Final Values) = .11

ADVERSE EVENTS:
Time Frame: Subjects were observed for 2.5 to 3 hours during the course of each of the three scanning sessions.
Groups:
- Methlyphenidate: 40mg methylphenidate
- Naltrexone: 40mg Naltrexone
- Placebo: Placebo
Arm/Group | Methlyphenidate | Naltrexone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes